CLINICAL TRIAL: NCT05724446
Title: A Phase 3, Multicenter, Randomized, Evaluator-blinded Clinical Trial to Assess the Safety and Efficacy of Clobetasol Propionate Ophthalmic Nanoemulsion, 0.05% Compared to Prednisolone Acetate, 1% in the Treatment of Inflammation After Cataract Surgery in Pediatric Population 0 to 3 Years of Age (CLOSE-3)
Brief Title: Clobetasol Propionate Ophthalmic Nanoemulsion, 0.05% in the Treatment of Inflammation After Cataract Surgery in Pediatric Population
Acronym: CLOSE-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Salvat (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLOBOF3-17IA03
Record Dates: First submitted 2023-01-23; First posted 2023-02-13 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Cataracts Infantile
Keywords: Cataract surgery; Inflammation; Pain
MeSH Terms: conditions — Inflammation; Pain | interventions — Clobetasol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clobetasol propionate (Experimental): One drop of Clobetasol propionate ophthalmic nanoemulsion, 0.05% will be administered of the study eye QID beginning the day after surgery (Day 1) for 14 days followed by a tapering period of 14 days.
  Interventions: Drug: Clobetasol Propionate
- Prednisolone acetate (Active Comparator): One drop of Prednisolone ophthalmic suspension, 1% will be administered of the study eye QID beginning the day after surgery (Day 1) for 14 days followed by a tapering period of 14 days.
  Interventions: Drug: Prednisolone acetate ophthalmic suspension, 1%

INTERVENTIONS:
Drug: Clobetasol Propionate — Clobetasol propionate ophthalmic nanoemulsion 0.05 % is an oil-in-water (O/W), clear or slightly yellowish nanoemulsion containing the active ingredient clobetasol propionate at a concentration of 0.05% weight per weight (w/w).
  Other Names: SVT-15473
  Arms: Clobetasol propionate
Drug: Prednisolone acetate ophthalmic suspension, 1% — Microfine sterile ophthalmic suspension of dense and whitish appearance.
  Arms: Prednisolone acetate

SUMMARY:
Multicenter, randomized, evaluator-blinded clinical trial compared to Prednisolone acetate, 1% in the treatment of inflammation and pain after cataract surgery in pediatric population. This study will assess the safety of Clobetasol propionate ophthalmic nanoemulsion, 0.05% to that of Prednisolone acetate, 1% when administering one drop four times a day (QID) for 14 days followed by a tapering period of 14 days after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 0 to 3 years old (have not had their 4th birthday) on the day of consent.
* Patients who are candidate for routine, uncomplicated cataract surgery in one eye with or without intraocular lens.
* Patients whose caregiver(s) is/are able and willing to comply with all treatment and follow-up procedures.
* Signed informed consent from (ICF) parents or patient's legally authorized representative(s).
* Patients who have undergone routine, uncomplicated cataract surgery in one eye with or without intraocular lens.
* Patients with clinical evidence of postoperative inflammation (anterior chamber inflammation grade > 0).

Exclusion Criteria:

* Presence of any active or suspected viral, bacterial, or fungal disease in the study eye.
* Active uveitis in the study eye.
* Ocular neoplasia in the study eye.
* Post-traumatic cataract in the study eye.
* Suspected permanent low vision or blindness in the fellow non-study eye. The study eye must not be the patient's only good eye.
* Use of any topical medication in the study eye within 2 days prior to surgery, except for those required for ocular examination or preoperative preparation.
* Systemic administration of any steroidal anti inflammatory drugs in the previous 2 weeks prior to the surgery.
* Systemic administration of any non-steroidal anti inflammatory drugs in the previous 48 hours prior to the surgery.
* Patient or patient's breastfeeding mother who is expected to use corticosteroids (except corticosteroid inhalers and dermatological corticosteroids, as long as they are not used on the eyelids or surrounding area, and oral prednisolone steaglate drops as part of the standard treatment after cataract surgery) or immunosuppressants during the 30 days following cataract surgery.
* History of steroid-induced increase in IOP in either eye.
* Patients with glaucoma, ocular hypertension, or those receiving IOP lowering therapy in either eye or systemically.
* Any current corneal abrasion or ulceration.
* Known or suspected allergy or hypersensitivity to similar drugs, such as other corticosteroids, or their components.
* Patients who have had ocular surgery in the study eye within 90 days prior to surgery.
* History of post-operative unresolved inflammation in the contralateral eye.
* Presence or history of chronic generalized systemic disease that the Investigator believes may either increase the risk to the subject or confound the results of the study (e.g., Diabetes mellitus, human immunodeficiency virus [HIV], acquired immunodeficiency syndrome [AIDS]).
* Any concurrent process which, in the opinion of the investigator, could impair patients' safety or limit adherence to the study protocol.
* Participation in any study of an investigational topical or systemic new drug or device within 30 days prior to screening, or at any time during the study.
* Prior participation in the study described in this protocol unless the patient wasn't randomized.

Ages: 0 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the safety of Clobetasol propionate ophthalmic nanoemulsion, 0.05% treatment after cataract surgery in pediatric population 0 to 3 years of age, compared to Prednisolone acetate ophthalmic suspension, 1%. | Day 43
  Number, frequency, severity, and relationship to IMP of adverse events (AEs) up to last study visit.

SECONDARY OUTCOMES:
Assess the efficacy on ocular inflammation of Clobetasol propionate ophthalmic nanoemulsion, 0.05% treatment after cataract surgery in pediatric population 0 to 3 years of age, compared to Prednisolone acetate ophthalmic suspension, 1%. | Day 15
  Percentage of patients with anterior chamber inflammation of grade 0. Anterior chamber inflammation is graded on a 5-point scale:
  0 = None: Clear anterior chamber with no visible clouding (Tyndall effect and cells combined). Red reflex normal.
  1. = Mild: Mild anterior chamber clouding. Clear iris pattern on visualization. Red reflex normal.
  2. = Moderate: Moderate anterior chamber clouding.
  3. = Severe: Severe anterior chamber clouding. Iris pattern not clearly visualized. Red reflex diminished.
  4. = Very severe: Severe anterior chamber clouding with a white and/or milky appearance of the anterior chamber. Red reflex absent or severely diminished.
Assess the efficacy on pain of Clobetasol propionate ophthalmic nanoemulsion, 0.05% treatment after cataract surgery in pediatric population 0 to 3 years of age, compared to Prednisolone acetate ophthalmic suspension, 1%. | Day 15
  Change in the Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Scale Score. Higher scores mean a worse outcome.
  Each of the five categories (F) Face; (L) Legs; (A) Activity; (C) Cry; (C) Consolability is scored from 0-2, which results in a total score between zero and ten.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospìtal Sant Joan de Deu, Barcelona, Spain